CLINICAL TRIAL: NCT00204217
Title: Monitoring of Intubation and Ventilation During Resuscitation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Oslo (Other)
Collaborators: Laerdal Medical (Industry); Ullevaal University Hospital (Other); Health Region East, Norway (Other); Norwegian Air Ambulance Foundation (Other); University of Stavanger (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 313-04124
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2007-08-27 (Estimated); Status verified 2007-08

CONDITIONS: Cardiac Arrest
Keywords: cardiac arrest; resuscitation; ventilation; impedance
MeSH Terms: conditions — Heart Arrest; Respiratory Aspiration | interventions — Intubation, Intratracheal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: endotracheal intubation

SUMMARY:
Airway control and ventilation is vital during cardiopulmonary resuscitation (CPR) in cardiac arrest. Endotracheal intubation is the gold standard for airway control, but several studies have shown high rates of unrecognized placements of the tube in the esophagus instead of in the airway out-of-hospital. This is lethal. There are no failproof technique for recognising such mistakes clinically in the cardiac arrest situation. Changes on the air volume in the lungs with ventilation changes the impedance (resistance to alternating current) through the thorax. This impedance is already measured routinely by the defibrillators used during CPR. We propose that we can measure ventilation volumes and also discover failed intubations by monitoring this impedance during CPR with the possibility of giving feedback on both to the rescuers.

DETAILED DESCRIPTION:
On the anesthesiologist manned ambulance in Oslo ventilation volumes during CPR will be controlled with a ventilator, the tidal volume varied in random order between 500, 700 and 100 ml, and the volumes be measured continuously as will the impedance between the defibrillator electrodes. In case of failed CPR, the patient will be declared dead. Thereafter the lungs will be ventilated with 700 ml followed by removal of the endotracheal tube, placement of an endotracheal tube in the esophagus and ventilation of this tube, again with monitoring of the impedance.

ELIGIBILITY:
Inclusion Criteria:

* Cardiac arrest

Exclusion Criteria:

* <18 years old trauma pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15
Dates: Start 2004-09; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
sensitivity/specificity for lung ventilation detection
correlation ventilation volume - impedance change

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Dorph, Principal Investigator — Ulleval University Hospital, University of Oslo
Locations (1):
- Ulleval University Hospital, Oslo, Norway